CLINICAL TRIAL: NCT04190381
Title: A Single-arm, Open Label, Single Center Study to Evaluate the Safety and Clinical Outcome of Using FR-Mask in Breast Cancer Patients With Radiation-irritated Skin After Radiotherapy
Brief Title: A Study to Evaluate the Safety and Clinical Outcome of Using FR-Mask in Breast Cancer Patients With Radiation-irritated Skin After Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chun Lin, Attending Physician, Division of Radiation Oncology, Principal Investigator, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH108-REC3-090
Record Dates: First submitted 2019-11-18; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
Keywords: deer antler velvet; radiation-irritated skin
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FR-Mask application (Experimental)
  Interventions: Other: FR-Mask

INTERVENTIONS:
Other: FR-Mask — The investigational medical product of this study is a biomedical repair mask, FR-MASK, acting like moisturizing lotion applied on breasts.
  The FR-Mask is applied to users' radiation-irritated breast skin for 15 to 20 minutes every 3 days.

SUMMARY:
The breast radiotherapy after breast-conserving surgery reduces the risk of recurrence and death and is widely used for standard treatment for breast cancer. However, radiation dermatitis is a major adverse event of breast radiotherapy. Radiation-irritated skin is a treatment-induced symptom caused by radiation dose-limiting toxicity. It damages skin structure and causes a variety of symptoms of cuticle thinning, sweat glands damage, sebaceous glands damage and basal membrane damage. Radiation-irritated skin also leads to lost work productivity, wound care costs, social isolation and altered body image. Thus, radiation-irritated skin can greatly impact the quality of life.

Several studies have examined the effects of numerous topical agents to reduce the dryness of skin. However, the reported results have not been clinically significant. Previous studies have shown that deer antler velvet extract possess inflammatory function and repair damaged follicles, sweat glands and sebaceous gland. And biocellulose membrane is a highly efficient media to introduce velvet extract to damaged skin tissue.

In this study, velvet extract combined with biocellolose membrane will be used in breast cancer patients to test the safety and efficacy to alleviate their radiation-irritated skin symptoms.

The investigational medical product of this study is a biomedical repair mask, FR-MASK ;the formula of FR-Mask is deer antler velvet, which is a traditional Chinese tonic medicine combined with high-adhesion biocellulose membrane.

The primary objective of this study is to test the safety and clinical outcomes of FR-Mask application in breast cancer patients who have radiation-irritated skin due to the post-operative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or non-pregnant females at least 20 years of age.
* Diagnosis of, non-inflammatory breast adenocarcinoma or in situ breast cancer and completed post-operative radiotherapy without concurrent chemotherapy.
* Breast adenocarcinoma previously treated by unilateral lumpectomy with or without adjuvant or neoadjuvant chemotherapy or hormonal treatment.
* Patients were scheduled to receive at least three sessions of radiotherapy per week (1 session per day) for at least five weeks using standard irradiation fraction (with at least 1.8 Gy per session) for total dose of at least 45 Gy.
* A time period of at least two weeks after radiotherapy before beginning the study.
* Participant must give informed consent.

Exclusion Criteria:

* Bilateral breast cancer
* Previous radiotherapy to the chest
* Chemotherapy concurrent with radiation treatment
* Prior breast reconstructions, implants, and/or expanders
* Known radiosensitivity syndromes (e.g. Ataxia-telangiectasia)
* Collagen vascular disease, vasculitis, unhealed surgical sites, breast infections or systemic lupus erythematosus (SLE)
* Participation in any clinical trial in the prior 30 days from baseline.
* Any condition that, in the judgement of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-06 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The change of scores of study questionnaire between baseline and each time point used to evaluate the breast cosmetic domain and specific breast pain domain. | Treatment: Day1, Day29, Day 57, Day85 and Post-treatment: 1 month
  Breast Cancer Treatment Outcome: Scale 1 = no difference between treated and untreated breast and area; 2 = slight difference between treated and untreated breast and area; 3 = moderate difference between treated and untreated breast and area; 4 = large difference between treated and untreated breast and area

SECONDARY OUTCOMES:
The change of moisture(water) percentage between baseline and each time point measured by skin analyzer (skin observed system) and skin checker (by electrical conductivity). | Treatment: Day1, Day29, Day 57, Day85 and Post-treatment: 1 month
The change of oil percentage between baseline and each time point measured by skin analyzer (skin observed system) and skin checker (by electrical conductivity). | Treatment: Day1, Day29, Day 57, Day85 and Post-treatment: 1 month
The change of pigment percentage between baseline and each time point measured by skin analyzer (skin observed system). | Treatment: Day1, Day29, Day 57, Day85 and Post-treatment: 1 month
The change of sensitivity percentage between baseline and each time point measured by skin analyzer (skin observed system). | Treatment: Day1, Day29, Day 57, Day85 and Post-treatment: 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen X, Wang Y, Wu Y, Wang L, Li W. [Protective effects of peptides from velvet antler of Cervus nippon on acute ischemic myocardial injury in rats]. Zhongguo Zhong Yao Za Zhi. 2009 Aug;34(15):1971-4. Chinese. PMID 19894547
- [Background] Suh JS, Eun JS, So JN, Seo JT, Jhon GJ. Phagocytic activity of ethyl alcohol fraction of deer antler in murine peritoneal macrophage. Biol Pharm Bull. 1999 Sep;22(9):932-5. doi: 10.1248/bpb.22.932. PMID 10513615
- [Background] Kim KS, Choi YH, Kim KH, Lee YC, Kim CH, Moon SH, Kang SG, Park YG. Protective and anti-arthritic effects of deer antler aqua-acupuncture (DAA), inhibiting dihydroorotate dehydrogenase, on phosphate ions-mediated chondrocyte apoptosis and rat collagen-induced arthritis. Int Immunopharmacol. 2004 Jul;4(7):963-73. doi: 10.1016/j.intimp.2004.04.010. PMID 15182735
- [Background] Fraser A, Haines SR, Stuart EC, Scandlyn MJ, Alexander A, Somers-Edgar TJ, Rosengren RJ. Deer velvet supplementation decreases the grade and metastasis of azoxymethane-induced colon cancer in the male rat. Food Chem Toxicol. 2010 May;48(5):1288-92. doi: 10.1016/j.fct.2010.02.024. Epub 2010 Feb 20. PMID 20176070
- [Background] Kuo CY, Wang T, Dai TY, Wang CH, Chen KN, Chen YP, Chen MJ. Effect of the Velvet Antler of Formosan Sambar Deer (Cervus unicolor swinhoei) on the Prevention of an Allergic Airway Response in Mice. Evid Based Complement Alternat Med. 2012;2012:481318. doi: 10.1155/2012/481318. Epub 2012 Dec 23. PMID 23346203